CLINICAL TRIAL: NCT04270955
Title: A Single Center Randomized Control Trial to Evaluate the Efficacy of Middle Meningeal Artery Embolization in the Treatment of Chronic Subdural Hematomas
Brief Title: Dartmouth Middle Meningeal Embolization Trial (DaMMET)
Acronym: DAMMET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Clifford J. Eskey, Director, Interventional Neuroradiology, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D20037
Record Dates: First submitted 2020-02-08; First posted 2020-02-17 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Chronic Subdural Hematoma; Subdural Hematoma
Keywords: Subdural Hematoma; Chronic Subdural Hematoma; Intracranial Hemorrhage
MeSH Terms: conditions — Hematoma, Subdural, Chronic; Hematoma, Subdural; Intracranial Hemorrhages

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Symptomatic, standard of care (Active Comparator): Patients in this group will be offered all procedures and care deemed appropriate by the Neurosurgeon in charge of their care. This could include surgical intervention, observation, medical management.
  Interventions: Procedure: Standard of care including possible surgical evacuation of subdural hematoma
- Symptomatic, MMA embolization + standard of care (Experimental): Patients in this group will be treated with the standard of care treatment (the same care described in the arm "Symptomatic, standard of care") but will also undergo MMA embolization of the affected side(s).
  Interventions: Procedure: Embolization of the Middle Meningeal Artery; Procedure: Standard of care including possible surgical evacuation of subdural hematoma
- Asymptomatic, standard of care (Active Comparator): Patients in this group will be offered all procedures deemed appropriate by the Neurosurgeon in charge of their care. This could include surgical intervention, observation, medical management.
  Interventions: Procedure: Standard of care including possible surgical evacuation of subdural hematoma
- Asymptomatic, standard of care + MMA embolization (Experimental): Patients in this group will be treated with the standard of care treatment (the same care described in the arm "Asymptomatic, standard of care") but will also undergo MMA embolization of the affected side(s).
  Interventions: Procedure: Embolization of the Middle Meningeal Artery; Procedure: Standard of care including possible surgical evacuation of subdural hematoma

INTERVENTIONS:
Procedure: Embolization of the Middle Meningeal Artery — Using established endovascular techniques and materials patient will have a diagnostic catheter based angiogram performed on the side(s) of the brain where the subdural hematoma is present. After verifying the vascular anatomy to ensure safety of the procedure the Middle Meningeal Artery will be embolized.
  Arms: Asymptomatic, standard of care + MMA embolization; Symptomatic, MMA embolization + standard of care
Procedure: Standard of care including possible surgical evacuation of subdural hematoma — Standard of care could include observation or intervention including surgical drainage of subdural hematoma by bedside drain, Subdural Evacuating Port System (SEPS), burr hole or craniotomy

SUMMARY:
Chronic subdural hematomas (cSDH) are one form of bleeding in the head. They are one of the most common diseases encountered by neurosurgeons across the country. The cSDH can push on the brain and produce symptoms that include seizures, weakness, loss of sensation, and confusion. Many of these cSDH produce repetitive bleeding.

Treatment has largely consisted of surgical drainage of hematoma (also known as a blood clot) through either a small hole in the skull or open surgery. However, it is common for the cSDH to reappear despite these procedures. A recent study has shown a treatment failure rate of 27% and a need for additional surgery at 19%.

A new approach to treatment of cSDH blocks the blood supply to the tissue that produces the repeated bleeding. Catheters are used to gain access to the middle meningeal artery (MMA), an artery that supplies the coverings of the brain. The artery is blocked using small particles or glue in a process called embolization. A recent pilot study of 72 patients who underwent MMA embolization showed a much lower rate of repeated bleeding. Based on these results, it is thought that this procedure holds promise in reducing the number of cSDH that require one or more operations. The goal of this study is to systematically examine if blocking the blood supply to the tissue responsible for repeated bleeding helps the cSDH resolve and improves patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Have radiographic imaging showing a cSDH > 7mm in maximal thickness encompassing > 50% of the convexity (non-focal).
* Capable of giving consent for the procedure or have an acceptable surrogate capable of giving consent on the subject's behalf

Exclusion Criteria:

* The cSDH is secondary to an underlying vascular malformation, tumor, cyst, spontaneous cerebrospinal fluid hypotension or previous craniotomy
* Life expectancy < 6 months
* Vascular anatomy that puts the patient at high risk for adverse events (e.g. critical carotid stenosis, abnormal external-internal carotid circulation)
* Incapable of being reasonably expected to be able to attend follow-up appointments at Dartmouth-Hitchcock Medical Center
* Vulnerable patients including homeless patients, incarcerated patients and mentally ill patients without appropriate medical decision-making proxy that the physician believes are incapable of appropriately assessing the risks of the procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-03-11 (Actual); Primary Completion 2024-01-11 (Actual); Study Completion 2024-01-11 (Actual)

PRIMARY OUTCOMES:
Radiographic resolution of hematoma | 3 months post-procedure
  CT scan to evaluate for residual hematoma, comparing baseline to 3 months
Radiographic resolution of hematoma | 6 months post-procedure
  CT scan to evaluate for residual hematoma, comparing baseline to 6 months. Can be canceled if cSDH is completely resolved at 3 months
Radiographic resolution of hematoma | 12 months post-procedure
  CT scan to evaluate for residual hematoma, comparing baseline to 12 months. Can be canceled if cSDH is completely resolved at 3 or 6 months

SECONDARY OUTCOMES:
Symptomatic improvement | 3 month follow up appointment
  HPI and neurologic exam (standard clinic follow-up) to compare to presenting symptoms.
Symptomatic improvement | 6 month follow up appointment
  HPI and neurologic exam (standard clinic follow-up) to compare to presenting symptoms. This may be canceled if the symptoms and hematoma are completely resolved at 3 months
Symptomatic improvement | 12 month follow up appointment
  HPI and neurologic exam (standard clinic follow-up) to compare to presenting symptoms. This may be canceled if the symptoms and hematoma are completely resolved at 3 or 6 months
NIH Stroke Scale | 3 months
  Comparison of NIHSS at admission to 3 month follow-up
NIH Stroke Scale | 6 months
  Comparison of NIHSS at admission to 6 month follow-up. May be canceled if cSDH resolved by 3 month follow up
NIH Stroke Scale | 6 months
  Comparison of NIHSS at admission to 12 month follow-up. May be canceled if cSDH resolved by 3 or 6 month follow up

CONTACTS AND LOCATIONS:
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No
There are no plans to share IPD at this time.